CLINICAL TRIAL: NCT01380145
Title: Pilot Study of recMAGE-A3 + AS15 ASCI as Consolidation for Multiple Myeloma Patients Undergoing Autologous Stem Cell Transplantation
Brief Title: MAGE-A3 Protein + AS15 as Consolidation for Multiple Myeloma Patients Undergoing Autologous Stem Cell Transplantation
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Ludwig Institute for Cancer Research (Other)
Collaborators: GlaxoSmithKline (Industry); MOUNT SINAI HOSPITAL (Other); NYU Langone Health (Other); Fox Chase Cancer Center (Other); Memorial Sloan Kettering Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LGS 2009-005; 10-051 (Other: Fox Chase Cancer Center); 10-216 (Other: Memorial Sloan-Kettering Cancer Center)
Record Dates: First submitted 2011-06-20; First posted 2011-06-27 (Estimated); Results first posted 2016-12-22 (Estimated); Last update posted 2022-10-25 (Actual); Status verified 2022-10

CONDITIONS: Multiple Myeloma
Keywords: multiple myeloma; MAGE-A3; autologous stem cell transplant
MeSH Terms: conditions — Multiple Myeloma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- recMAGE-A3 Protein + AS15 Adjuvant (Experimental): Subjects received a total of 8 pre- and post-auto-SCT immunizations with recMAGE-A3 + AS15.
  Interventions: Biological: recMAGE-A3 Protein + AS15 Adjuvant

INTERVENTIONS:
Biological: recMAGE-A3 Protein + AS15 Adjuvant — recMAGE-A3 + AS15 was administered intramuscularly at a dose of 300 µg recMAGE-A3, with no dose adjustments permitted. The first immunization was administered 6 to 15 week prior to auto-SCT, with subsequent immunizations administered on Days 10, 31, 52, 73, and 94 (± 3 days) and Days 180 and 270 (± 7 days) after auto-SCT.
  Other Names: Antigen-specific cancer immunotherapeutic (ASCI)

SUMMARY:
This was an open-label, single-arm, pilot study of the recombinant MAGE-A3 protein plus the immunological adjuvant AS15 (recMAGE-A3 + AS15) in subjects with symptomatic multiple myeloma who had completed induction therapy with at least a Very Good Partial Response (VGPR) by the International Myeloma Working Group (IMWG) criteria and who were eligible for high-dose chemotherapy with autologous stem cell transplant (auto-SCT). The primary objective was to determine the safety and tolerability of immunizations when administered prior to stem cell mobilization and multiple times after stem cell reinfusion. Secondary objectives were to assess the humoral and cellular immunogenicity and clinical outcomes of immunization.

DETAILED DESCRIPTION:
Subjects were enrolled sequentially following confirmation of eligibility criteria, including International Staging System (ISS) stage 1, 2, or 3 multiple myeloma with MAGE-A3 tumor antigen expression. Subjects received a total of 8 immunizations with 300 µg of recMAGE-A3 + AS15. The first immunization was administered approximately 6 to 15 weeks prior to auto-SCT (Day 0), with subsequent immunizations administered every 3 weeks (± 3 days) starting 10 days after auto-SCT (ie, Days 10, 31, 52, 73, and 94). Two additional immunizations were administered at 3-month intervals (± 7 days, ie, Days 180 and 270). No dose adjustments were allowed. Platelet counts must have been ≥ 50 x 10E9/L prior to immunization, with blood product transfusions permitted as necessary.

The process for auto-SCT comprised the following: (1) up to 3 steady-state leukopheresis procedures to collect and freeze a sufficient quantity of peripheral blood mononuclear cells (PBMCs), with the first leukopheresis performed 3 weeks (± 6 days) after the first immunization; (2) stem cell mobilization with cyclophosphamide, granulocyte-colony stimulating factor (G-CSF) and/or plerixafor; (3) high-dose melphalan (total dose 200 mg/m2) on Days -3 through -1; (4) auto-SCT on Day 0; and (5) re-infusion with thawed PBMCs on Day 3.

ELIGIBILITY:
Inclusion Criteria:

1. Symptomatic multiple myeloma, ISS stage 1, 2 or 3 within 12 months of starting therapy.
2. Completion of induction therapy with VGPR, or better, by IMWG criteria. All induction myeloma therapy (oral or intravenous, including steroids) must have been discontinued for 3 weeks prior to the first immunization. Subjects did not need to have measurable disease at the time of the screening visit.
3. Signed separate informed consent for stem cell mobilization and high-dose chemotherapy/auto-SCT, and was found to be eligible for SCT by standard institutional criteria.
4. MAGE-A3 expression determined by immunohistochemistry (IHC) present in a bone marrow specimen or plasmacytoma specimen.
5. Eastern Cooperative Oncology Group (ECOG) performance status 0 to 1.
6. The following laboratory parameters within the ranges specified:

   * Neutrophil count: ≥ 1.5 x 109/L
   * Lymphocyte count: ≥ 0.5 x 109/L
   * Platelet count: ≥ 50 x 109/L
   * Serum creatinine: ≤ 2 mg/dL
   * Serum bilirubin: < 1.5 x the upper limit of normal (ULN)
   * Aspartate and alanine aminotransferase (AST and ALT): < 2 x ULN
   * Hemoglobin: ≥ 8.0 g/dL
   * International normalized ratio (INR): ≤ 1.5
   * Partial thromboplastin time: ≤ 1.5 x ULN (unless known history of anti-phospholipid antibody or lupus anticoagulant)
7. Age ≥ 18 years.
8. Able and willing to give valid written informed consent.

Exclusion Criteria:

1. Prior treatment with melphalan (Alkeran®), other than 1 cycle (4 days) of oral melphalan.
2. Prior autologous or allogeneic SCT.
3. Prior immunization against MAGE-A3 or other cancer-testis antigens.
4. Concurrent malignancies, except for treated non-melanoma skin cancer and cervical carcinoma in situ.
5. Known immunodeficiency, human immunodeficiency virus (HIV) positivity, or active hepatitis B or C.
6. Known allergy or history of life-threatening reaction to G-CSF or GM-CSF.
7. History of autoimmune disease (eg., rheumatoid arthritis, lupus), other than vitiligo, diabetes, or treated thyroiditis.
8. History of severe allergic reactions to vaccines or unknown allergens.
9. History of myocardial infarction, angina, congestive heart failure, ventricular tachyarrhythmia, stroke or transient ischemic attack within the previous 6 months.
10. Other serious illnesses or co-morbid conditions (e.g., serious infections requiring antibiotics, bleeding disorders, other heart or lung conditions) that, in the opinion of the investigator, made the subject inappropriate for high-dose melphalan and auto-SCT.
11. Pregnancy and breastfeeding.
12. Participation in any other clinical trial involving another investigational agent within 4 weeks prior to first immunization.
13. Mental impairment that may have compromised the ability to give informed consent and comply with the requirements of the study.
14. Lack of availability for immunological and clinical follow-up assessments.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2011-09; Primary Completion 2014-07 (Actual); Study Completion 2014-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Hearn J Cho, MD, PhD, Study Chair — MOUNT SINAI HOSPITAL; Michael Millenson, MD, Principal Investigator — Fox Chase Cancer Center; Nikoletta Lendvai, MD, PhD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (4):
- United States (4):
  - New York University School of Medicine, New York, New York
  - Mount Sinai Hospital, New York, New York
  - Memorial Sloan-Kettering Cancer Center, New York, New York
  - Fox Chase Cancer Center, Philadelphia, Pennsylvania

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Cohen AD, Lendvai N, Nataraj S, Imai N, Jungbluth AA, Tsakos I, Rahman A, Mei AH, Singh H, Zarychta K, Kim-Schulze S, Park A, Venhaus R, Alpaugh K, Gnjatic S, Cho HJ. Autologous Lymphocyte Infusion Supports Tumor Antigen Vaccine-Induced Immunity in Autologous Stem Cell Transplant for Multiple Myeloma. Cancer Immunol Res. 2019 Apr;7(4):658-669. doi: 10.1158/2326-6066.CIR-18-0198. Epub 2019 Feb 11. PMID 30745365

RESULTS

PARTICIPANT FLOW:
Groups:
- All Enrolled Subjects: Subjects received a total of 8 pre- and post-auto-SCT immunizations with recMAGE-A3 + AS15 administered intramuscularly at a dose of 300 µg recMAGE-A3, with no dose adjustments permitted. The first immunization was administered 6 to 15 week prior to auto-SCT, with subsequent immunizations administered on Days 10, 31, 52, 73, and 94 (± 3 days) and Days 180 and 270 (± 7 days) after auto-SCT.
Period: Overall Study
Arm/Group | All Enrolled Subjects
Started | 13
Completed | 9
Not Completed | 4
Not completed — Progressive disease | 4

BASELINE CHARACTERISTICS:
Population: Includes all subjects enrolled in the study.
Groups:
- All Enrolled Subjects: Includes all subjects enrolled in the study.
Arm/Group | All Enrolled Subjects
Number analyzed (Participants) | 13
Age, Continuous [Mean (Standard Deviation); unit: years] | 54.3 (10.33)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4
  Male | 9
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 12
  Unknown or Not Reported | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 2
  White | 10
  More than one race | 0
  Unknown or Not Reported | 1
Region of Enrollment [Number; unit: participants]
  United States | 13
Body Mass Index [Mean (Standard Deviation); unit: kg/m^2] | 30.2 (4.74)
Response to Prior Induction Therapy [Number; unit: participants] — Complete Response (CR): negative immunofixation on serum/urine, disappearance of soft tissue plasmacytomas, <5% plasma cells in bone marrow
  Stringent CR (sCR): CR + normal free light chain (FLC) ratio and absence of clonal cells in bone marrow
  Very Good Partial Response (VGPR): Serum/urine M-component detectable by immunofixation but not electropheresis OR ≥90% reduction in serum M-component + urine M-component <100 mg/24 hrs
  PR: ≥50% reduction of serum M-protein and reduction in 24-hr urinary M-protein by ≥90% or to <200 mg/24 hrs
  Stable disease: not response or progression
  participants
    Complete Response | 1
    Very Good Partial Response | 12

OUTCOME MEASURES:

1. Primary Outcome: Assessment of Safety of recMAGE-A3 + AS15
Description: Analysis of treatment-emergent adverse events (TEAEs) reported from clinical laboratory tests, physical examinations, and vital signs, with severity graded according to the NCI CTCAE, Version 4.0.
Time Frame: Continuously for up to 14 months
Population: The Safety Analysis Set comprises all subjects who received at least 1 immunization with study drug.
Measure: Number; unit: participants
Groups:
- Safety Analysis Set: Includes all subjects who received at least 1 immunization with study drug.
Arm/Group | Safety Analysis Set
Number analyzed (Participants) | 13
participants
  Any TEAE | 13
  Grade 3 TEAE | 8
  Grade 4 TEAE | 4
  Grade 5 TEAE (Death) | 0
  Treatment-related TEAE | 10
  SAE | 4
  TEAE leading to withdrawal | 0

2. Secondary Outcome: Induction or Augmentation of MAGE-A3-Specific Humoral Immunity
Description: Humoral immunity was determined by enzyme-linked immunosorbent assay (ELISA) to measure the presence of circulating antibodies to MAGE-A3. Titers against an antigen were considered significant if they were >100. Induction of responses was considered significant if there was a change from undetectable (<100) to detectable (>100) or if there was an at least 4-fold increase in titers over time.
Time Frame: Baseline, first immunization, and first and second leukopheresis prior to auto-SCT; Days 31, 73, 194, 284, and 374 after auto-SCT
Population: The Immunogenicity Analysis Set comprises all subjects who received at least 1 immunization with study drug and had a baseline and at least 1 post-baseline immunity assessment.
Measure: Number; unit: participants
Groups:
- Immunogenicity Analysis Set: Includes all subjects who received at least 1 immunization with study drug and had a baseline and at least 1 post-baseline immunity assessment.
Arm/Group | Immunogenicity Analysis Set
Number analyzed (Participants) | 13
participants
  Seroconversion after 1 immunization | 3
  Seroconversion after 2 immunizations | 8
  Seroconversion after 3-4 immunizations | 2

3. Secondary Outcome: Induction or Augmentation of MAGE-A3-Specific Cellular Immunity
Description: Cellular immunity was determined by enzyme-linked immunosorbent spot assay (ELISPOT) or intracellular flow cytometry to determine peripheral blood levels of interferon gamma-producing CD4+ and CD8+ T cells specific for MAGE-A3. Results were considered significant if > 50 spots and > 2 times the number of spots to negative control were observed.
Time Frame: as for outcome 2
Population: as for outcome 2
Measure: Number; unit: participants
Arm/Group | Immunogenicity Analysis Set
Number analyzed (Participants) | 13
participants
  Baseline CD4 T cell response | 6
  Post-immunization CD4 T-cell response/increase | 13
  Baseline CD8 T cell response | 0
  Post-immunization CD8 T-cell response/increase | 3

4. Secondary Outcome: Assessment of Tumor Response
Description: Tumor responses were evaluated using appropriate imaging methods and were categorized according to the IMWG criteria, which includes the following response designations:
  Complete Response (CR): negative immunofixation on serum/urine, disappearance of soft tissue plasmacytomas, <5% plasma cells in bone marrow; Stringent CR (sCR): CR + normal free light chain (FLC) ratio and absence of clonal cells in bone marrow; Very Good Partial Response (VGPR): Serum/urine M-component detectable by immunofixation but not electropheresis OR ≥90% reduction in serum M-component + urine M-component <100 mg/24 hrs; Partial Response (PR): ≥50% reduction of serum M-protein and reduction in 24-hr urinary M-protein by ≥90% or to <200 mg/24 hrs Stable disease: not response or progression
Time Frame: At 3 and 12 months after auto-SCT
Population: The Evaluable Analysis Set comprises all subjects who received at least 1 immunization with study drug and had a baseline and at least 1 post-baseline disease assessment.
Measure: Number; unit: participants
Groups:
- Evaluable Analysis Set: Includes all subjects who received at least 1 immunization with study drug and had a baseline and at least 1 post-baseline disease assessment.
Arm/Group | Evaluable Analysis Set
Number analyzed (Participants) | 13
participants
  Day 94: Stringent Complete Response | 2
  Day 94: Complete Response | 3
  Day 94: Very Good Partial Response | 8
  Day 360: Stringent Complete Response | 4
  Day 360: Complete Response | 1
  Day 360: Very Good Partial Response | 4
  Day 360: Progressive Disease | 4

5. Secondary Outcome: Assessment of Survival and Time to Subsequent Therapy
Description: Progression-free survival (PFS) was calculated as the date from first immunization to first observation of disease progression or death due to any cause, censored on the start date of subsequent therapy or at the last date of disease assessment for subjects without a PFS event. Overall survival (OS) was calculated as the date from first immunization to death due to any cause, censored at the date of last follow-up for subjects who were alive at the time of the analysis. Time to subsequent therapy was calculated as the date from first immunization to start of subsequent therapy for myeloma, censored at the date of death or last follow-up for subjects who did not receive subsequent therapy.
Time Frame: Continuously on study and for up to 5 years post-study
Population: as for outcome 4
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Evaluable Analysis Set
Number analyzed (Participants) | 13
days
  Median PFS using the Kaplan-Meier Method | 751 [379 to NA] — Upper limit of the confidence interval was not reached.
  Median OS using the Kaplan-Meier Method | 829 [829 to NA] — Upper limit of the confidence interval was not reached.
  Median Time to Subsequent Therapy using Kaplan-Meier Method | 805 [414 to NA] — Upper limit of the confidence interval was not reached.

ADVERSE EVENTS:
Time Frame: All AEs occurring between the date of enrollment and the off-study date (i.e., for up to 14 months) were documented, regardless of the causal relationship to study drug. AEs occurring or worsening after the first dose of study drug were considered treatment emergent (i.e., TEAEs).
Description: AE documentation included onset/resolution dates, severity using NCI CTCAE (v4.0), seriousness, study drug action taken, treatment, and outcome. In summaries, treatment-related AEs included those with a "possible", "probable", or "definite" relationship to study drug; preferred terms were counted only once per subject at the maximum reported grade.
Arm/Group | Safety Analysis Set
Serious Adverse Events (participants affected / at risk) | 4/13
Other Adverse Events (participants affected / at risk) | 13/13
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Safety Analysis Set (N=13)
Psoriasis (Skin and subcutaneous tissue disorders) | 1 (1) — Grade 2, unresolved; represents a potential immune-mediated disease (pIMD)
Connective tissue disorder (Musculoskeletal and connective tissue disorders) | 1 (1) — Grade 3, unresolved
Diarrhoea (Gastrointestinal disorders) | 1 (1) — Grade 3, resolved
Vomiting (Gastrointestinal disorders) | 1 (1) — Grade 2, resolved
Nausea (Gastrointestinal disorders) | 1 (1) — Grade 2, resolved
Injection site reaction (General disorders) | 1 (1) — Grade 1, resolved
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1) — Grade 2, resolved
Atrial fibrillation (Cardiac disorders) | 1 (1) — Grade 3, resolved
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1 (1) — Grade 3, resolved
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Safety Analysis Set (N=13)
Nausea (Gastrointestinal disorders) | 9
Fatigue (General disorders) | 8
Decreased appetite (Metabolism and nutrition disorders) | 7
Diarrhoea (Gastrointestinal disorders) | 6
Thrombocytopenia (Blood and lymphatic system disorders) | 6
Bone pain (Musculoskeletal and connective tissue disorders) | 5
Constipation (Gastrointestinal disorders) | 5
Headache (Nervous system disorders) | 5
Insomnia (Psychiatric disorders) | 5
Alopecia (Skin and subcutaneous tissue disorders) | 4
Anaemia (Blood and lymphatic system disorders) | 4
Febrile neutropenia (Blood and lymphatic system disorders) | 4
Hypokalaemia (Metabolism and nutrition disorders) | 4
Injection site reaction (General disorders) | 4
Injection site pain (General disorders) | 4
Mucosal inflammation (General disorders) | 4
Paraesthesia (Nervous system disorders) | 4
Pyrexia (General disorders) | 4
Abdominal pain (Gastrointestinal disorders) | 3
Anxiety (Psychiatric disorders) | 3
Flushing (Vascular disorders) | 3
Leukopenia (Blood and lymphatic system disorders) | 3
Neuropathy peripheral (Nervous system disorders) | 3
Rash (Skin and subcutaneous tissue disorders) | 3
Sinusitis (Infections and infestations) | 3
Upper respiratory tract infection (Infections and infestations) | 3
Urticaria (Skin and subcutaneous tissue disorders) | 3
Vomiting (Gastrointestinal disorders) | 3
Arthralgia (Musculoskeletal and connective tissue disorders) | 2
Chest discomfort (General disorders) | 2
Chills (General disorders) | 2
Cough (Respiratory, thoracic and mediastinal disorders) | 2
Dizziness (Nervous system disorders) | 2
Dyspepsia (Gastrointestinal disorders) | 2
Hypocalcaemia (Metabolism and nutrition disorders) | 2
Hypomagnesaemia (Metabolism and nutrition disorders) | 2
Influenza like illness (General disorders) | 2
Myalgia (Musculoskeletal and connective tissue disorders) | 2
Neutropenia (Blood and lymphatic system disorders) | 2
Oedema peripheral (General disorders) | 2
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 2
Acute sinusitis (Infections and infestations) | 1
Agitation (Psychiatric disorders) | 1
Back pain (Musculoskeletal and connective tissue disorders) | 1
Blood testosterone decreased (Investigations) | 1
Bronchitis (Infections and infestations) | 1
Diabetes mellitus (Metabolism and nutrition disorders) | 1
Drug hypersensitivity (Immune system disorders) | 1
Dry mouth (Gastrointestinal disorders) | 1
Dry skin (Skin and subcutaneous tissue disorders) | 1
Dysgeusia (Nervous system disorders) | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1
Fungal skin infection (Infections and infestations) | 1
Haematuria (Renal and urinary disorders) | 1
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1
Hypertension (Vascular disorders) | 1
Hypoalbuminaemia (Metabolism and nutrition disorders) | 1
Hypotension (Vascular disorders) | 1
Infection (Infections and infestations) | 1
Influenza (Infections and infestations) | 1
Infusion related reaction (General disorders) | 1
Ligament rupture (Injury, poisoning and procedural complications) | 1
Malaise (General disorders) | 1
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1
Nail discolouration (Skin and subcutaneous tissue disorders) | 1
Nodule (General disorders) | 1
Non-cardiac chest pain (General disorders) | 1
Oedema (General disorders) | 1
Oral pain (Gastrointestinal disorders) | 1
Orthostatic hypotension (Vascular disorders) | 1
Osteopenia (Musculoskeletal and connective tissue disorders) | 1
Peripheral sensory neuropathy (Nervous system disorders) | 1
Pharyngeal inflammation (Respiratory, thoracic and mediastinal disorders) | 1
Pneumonia (Infections and infestations) | 1
Proctalgia (Gastrointestinal disorders) | 1
Proctitis (Gastrointestinal disorders) | 1
Productive cough (Respiratory, thoracic and mediastinal disorders) | 1
Pruritus (Skin and subcutaneous tissue disorders) | 1
Pulmonary congestion (Respiratory, thoracic and mediastinal disorders) | 1
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 1
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 1
Skin papilloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Somnolence (Nervous system disorders) | 1
Stress fracture (Injury, poisoning and procedural complications) | 1
Syncope (Nervous system disorders) | 1
Urinary tract infection (Infections and infestations) | 1
Vaginal haemorrhage (Reproductive system and breast disorders) | 1
Vessel puncture site reaction (General disorders) | 1
Vitamin K deficiency (Metabolism and nutrition disorders) | 1
Vulvitis (Infections and infestations) | 1
Weight increased (Investigations) | 1
Ear disorder (Ear and labyrinth disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less